CLINICAL TRIAL: NCT05878093
Title: A Randomized, Double-blind, Placebo-controlled Efficacy and Safety Study of Dupilumab, in Chinese Adult Participants With Chronic Rhinosinusitis With Nasal Polyposis (CRSwNP) on a Background Therapy With Intranasal Corticosteroids
Brief Title: Dupilumab in Chinese Adult Participants With CRSwNP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17026; U1111-1256-9711 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — dupilumab; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): Dupilumab every 2 weeks (Q2W) via SC injection
  Interventions: Drug: Dupilumab; Drug: Budesonide
- Placebo (Placebo Comparator): Placebo matching dupilumab Q2W via SC injection
  Interventions: Drug: Placebo; Drug: Budesonide

INTERVENTIONS:
Drug: Dupilumab — solution for subcutaneous injection
  Arms: Dupilumab
Drug: Placebo — solution for subcutaneous injection
  Arms: Placebo
Drug: Budesonide — nasal spray (suspension)

SUMMARY:
This is a parallel group, Phase 3, 2-arm study for treatment. The purpose of this study is to evaluate dupilumab subcutaneous (SC) injections compared to placebo in Chinese adult participants with CRSwNP, on a background therapy with intranasal corticosteroids (budesonide nasal spray).

Study details include:

* The study duration will be up to 40 weeks.
* The treatment duration will be up to 24 weeks.
* The number of visits will be 7.

DETAILED DESCRIPTION:
up to 40 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of signing the informed consent
* Participants with bilateral sino-nasal polyposis that despite prior treatment with SCS anytime within the past 2 years; and/or who have a medical contraindication/intolerance to SCS; and/or had prior surgery for NP at Visit 1 have:

  1. An endoscopic bilateral NPS at Visit 1 of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity) as per central assessment
  2. Ongoing symptoms (for at least 8 weeks before Visit 1) of:

     * Nasal congestion/blockade/obstruction with moderate or severe symptom severity (Score 2 or 3) at Visit 1 and a weekly average severity of greater than 1 at time of randomization (Visit 2) AND
     * Another symptom such as loss of smell, rhinorrhea (anterior/posterior)

Note: Plan to enroll at least 85% (approximately 52) participants with CRSwNP meeting following criterion:

• Participants with peripheral blood eosinophil count ≥300/mm3

* Contraceptive use should be consistent with the regulations regarding the methods of contraception for those participating in clinical studies
* Capable of giving signed informed consent

Exclusion Criteria:

* Participants with conditions/concomitant diseases making them non-evaluable at Visit 1 or for the primary efficacy endpoint (ie, NPS)
* Participants with nasal cavity malignant tumor and benign tumors (eg, papilloma, hemangioma, etc)
* Participant with historical spirometry results which showed 50% or less of predicted normal of forced expiratory volume in one second (FEV1)
* Diagnosed with; suspected of, or at high risk of endoparasitic infection, and/or use of antiparasitic drug within 2 weeks before Visit 1 or during the screening period
* History of human immunodeficiency virus infection or positive HIV 1/2 serology at Visit 1
* Known or suspected immunodeficiency
* Participants with active Tuberculosis (TB), non-tuberculous mycobacterial infection or a history of incompletely treated TB will be excluded from the study unless it is well documented by a specialist that the participant has been adequately treated and can now start treatment with a biologic agent, in the medical judgment of the Investigator and/or infectious disease specialist. Tuberculosis testing will be performed according to local guidelines if required by regulatory authorities or ethics boards, or if TB is suspected by the investigator
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before Visit 1 or during the screening period
* Active malignancy or history of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix and completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin
* Known or suspected alcohol and/or drug abuse
* History of systemic hypersensitivity or anaphylaxis to dupilumab including any excipient
* Participants meet any contraindications or warning on product labeling for budesonide nasal spray
* Severe concomitant illness(es) that, in the Investigator's judgement, would adversely affect the participant's participation in the study.
* Participants with any other medical or psychological condition including relevant laboratory or electrocardiogram (ECG) abnormalities at screening that, in the opinion of the Investigator, suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study participant as a result of his/her participation in this clinical trial, may make participant's participation unreliable, or may interfere with study assessments. The specific justification for participants excluded under this criterion will be noted in study documents (chart notes, case report form (CRF), etc)
* Planned major surgical procedure during the participant's participation in this study
* Participants who have taken:

Biologic therapy/systemic immunosuppressant/immunomodulator within 4 weeks before Visit 1 or 5 half-lives, whichever is longer.

Any investigational monoclonal antibody (mAb) within 5 half-lives or within 6 months before Visit 1 if the half-life is unknown.

Anti-immunoglobulin E therapy (omalizumab) within 4 months prior to Visit 1.

* Treatment with a live (attenuated) vaccine within 4 weeks prior to Visit 1
* Participants who are receiving leukotriene antagonists/modifiers within 4 weeks before V1 or 5 half-lives, whichever is longer, unless patient is on a continuous treatment for at least 4 weeks before Visit 1
* Initiation of allergen immunotherapy within 3 months prior to Visit 1 or a plan to begin therapy or change its dose during the run-in or randomized treatment period
* Participants who have undergone any intranasal and/or sinus surgery (including polypectomy) within 6 months prior to Visit 1 or sino-nasal surgery changing the lateral wall structure of the nose making the evaluation of NPS impossible
* Use of any prohibited medications and procedures during screening period or planned use during screening or study treatment period
* Either intravenous immunoglobulin (IVIG) therapy and/or plasmapheresis within 4 weeks before Visit 1
* Current participation in any clinical trial of an investigational drug or device or participation within 3 months before V1 or 5 half-lives of the investigational compound, whichever is longer
* Participation in a prior dupilumab clinical study or have been treated with commercially available dupilumab
* Patients with any of the following result at the screening visit (Visit 1):

Positive (or indeterminate) hepatitis B surface antigen (HBsAg) or, Positive total Hepatitis B core antibody (HBc Ab) confirmed by positive hepatitis B virus (HBV) DNA or, Positive HCV Ab confirmed by positive hepatitis C Virus (HCV) RNA.

* noninvestigational medicinal product(NIMP) noncompliance at Visit 2 (<80%)
* Any condition that could make the participant noncompliant with the study procedures and daily assessment in the e-diary
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized.
* Participants not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560010, Chengdu
  - Investigational Site Number : 1560014, Chongqing
  - Investigational Site Number : 1560022, Fuzhou
  - Investigational Site Number : 1560012, Guangzhou
  - Investigational Site Number : 1560011, Guangzhou
  - Investigational Site Number : 1560004, Hangzhou
  - Investigational Site Number : 1560006, Hefei
  - Investigational Site Number : 1560016, Jinan
  - Investigational Site Number : 1560025, Jingzhou
  - Investigational Site Number : 1560013, Qingdao
  - Investigational Site Number : 1560017, Shanghai
  - Investigational Site Number : 1560018, Taiyuan
  - Investigational Site Number : 1560007, Wuhan
  - Investigational Site Number : 1560021, Wuhan
  - Investigational Site Number : 1560009, Yantai
  - Investigational Site Number : 1560020, Zibo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17026 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25260&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 centers in China. A total of 151 participants were screened from 16 May 2023 to 27 February 2024, of which 88 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 63 participants were randomized in a 1:1 ratio to receive either matching placebo or dupilumab. Randomization was stratified by screening blood eosinophil count (>=300 cells per cubic millimeter [/mm^3] or <300 cells/mm^3).
Groups:
- Placebo: Participants received placebo matched to dupilumab subcutaneous (SC) injection every 2 weeks (q2w) from Day 1 up to 24 weeks.
- Dupilumab 300 mg q2w: Participants received dupilumab 300 milligrams (mg) SC injection q2w from Day 1 up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w
Started | 32 | 31
Completed | 29 | 30
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants with a treatment kit number allocated and recorded in the interactive response technology database, regardless of whether the treatment kit was used or not.
Groups:
- Placebo: Participants received placebo matched to dupilumab SC injection q2w from Day 1 up to 24 weeks.
- Dupilumab 300 mg q2w: Participants received dupilumab 300 mg SC injection q2w from Day 1 up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.3) | 47.1 (12.1) | 48.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 32 | 31 | 63
Nasal Polyps Score (NPS) [Mean (Standard Deviation); unit: score on a scale] — NPS was sum of right and left nostril scores.For each nostril,NPS was graded based on polyp size,ranged from 0:no polyps,1:small polyps in middle meatus not reaching below inferior border of middle turbinate,2:polyps reaching below lower border of middle turbinate,3:large polyps reaching lower border of inferior turbinate or polyps medial to middle turbinate,4:large polyps causing complete obstruction of inferior nasal cavity.Total NPS:sum of right and left nostril scores;range:0(no polyps) to 8(large polyps).Higher scores:more severe disease.Baseline:last available value before randomization.
  score on a scale | 5.84 (1.60) | 5.53 (1.41) | 5.69 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Nasal Polyps Score at Week 24
Description: The NPS was the sum of the right and left nostril scores and assessed by central video recordings of bilateral nasal endoscopy. For each nostril, NPS was graded based on polyp size which ranged from 0: no polyps, 1: small polyps in the middle meatus not reaching below the inferior border of the middle turbinate, 2: polyps reaching below the lower border of the middle turbinate, 3: large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate, 4: large polyps causing complete obstruction of the inferior nasal cavity. Total NPS was the sum of right and left nostril scores; ranged from 0 (no polyps) to 8 (large polyps). Higher scores indicated more severe disease. Baseline was defined as the last available value before randomization.
Time Frame: Baseline (Day 1) and Week 24
Population: The intent-to-treat (ITT) population included all randomized participants analyzed according to the treatment group allocated by randomization, regardless of whether the treatment kit was used or not.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
score on a scale | -0.50 (0.30) | -2.34 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Test type: Superiority — A hierarchical procedure was used to control type I error and handle primary and first 4 secondary endpoints (reported sequentially) analyses at a 2-sided significance level of 0.05; p < 0.0001, ANCOVA; Least square mean difference = -1.84, 95% CI 2-sided [-2.53 to -1.15] — Data was analyzed by fitting an analysis of covariance (ANCOVA) model with the corresponding baseline value, treatment group, and screening blood eosinophil count strata as covariates

2. Secondary Outcome: Change From Baseline in Nasal Congestion/Obstruction Score (NCS) at Week 24
Description: The NCS was a patient reported outcome to evaluate nasal congestion/obstruction, a major clinical symptom in chronic rhinosinusitis phenotype with nasal polyps. The NCS was assessed by the participant on a daily basis from visit 1 and throughout the study. It consisted of a 0 to 3 categorical scale, where 0: no symptoms, 1: mild symptoms, 2: moderate symptoms and 3: severe symptoms. Higher scores indicated more severity. The Week 24 analysis score was calculated as the average of all scores during the 4 weeks before Week 24. Baseline was defined as the average of the scores in the 7 days prior to randomization.
Time Frame: Baseline (Day -7 to Day -1) and Week 24
Population: The ITT population included all randomized participants analyzed according to the treatment group allocated by randomization, regardless of whether the treatment kit was used or not.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
score on a scale | -0.52 (0.18) | -1.06 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0126, ANCOVA; Least square mean difference = -0.54, 95% CI 2-sided [-0.97 to -0.12] — Data was analyzed by fitting an ANCOVA model with the corresponding baseline value, treatment group, and screening blood eosinophil count strata as covariates

3. Secondary Outcome: Change From Baseline in Total Symptoms Score (TSS) at Week 24
Description: The TSS was a reflective score of the worst symptom severity over the past 24 hours by the participant. It was assessed by the participant on a daily basis from visit 1 and throughout the study. It consisted of the sum of the following rhinosinusitis symptom questions: nasal congestion, decreased/loss of sense of smell, rhinorrhea (average of anterior/posterior nasal discharge); each assessed on 0 to 3 categorical scale, where 0: no symptoms, 1: mild symptoms, 2: moderate symptoms and 3: severe symptoms. The TSS was a composite score by summing the above symptom scores and ranged from 0 (no symptoms) to 9 (severe symptoms). Higher scores indicated greater overall symptom severity. The Week 24 analysis score was calculated as the average of all scores during the 4 weeks before Week 24. Baseline was defined as the average of the scores in the 7 days prior to randomization.
Time Frame: Baseline (Day -7 to Day -1) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
score on a scale | -1.07 (0.43) | -2.75 (0.43)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0008, ANCOVA; Least square mean difference = -1.68, 95% CI 2-sided [-2.67 to -0.69] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in the Severity of Decreased/Loss of Smell at Week 24
Description: The decreased/loss of sense of smell severity was a reflective score of the worst symptom severity over the past 24 hours. It was assessed by the participant on a daily basis from visit 1 and throughout the study, using an e-diary. It consisted of a 0 to 3 categorical scale, where 0: no symptoms, 1: mild symptoms, 2: moderate symptoms and 3: severe symptoms. Higher scores indicated more severe symptoms. The Week 24 analysis score was calculated as the average of all scores during the 4 weeks before Week 24. Baseline was defined as the average of the scores in the 7 days prior to randomization.
Time Frame: Baseline (Day -7 to Day -1) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
score on a scale | -0.23 (0.20) | -0.86 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0072, ANCOVA; Least square mean difference = -0.62, 95% CI 2-sided [-1.08 to -0.17] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in Total Score of 22-Items Sinonasal Outcome Test (SNOT-22) at Week 24
Description: The SNOT-22 was a validated 22-items questionnaire to assess the impact of chronic rhinosinusitis on health-related quality of life (HRQoL) with a recall period of 2 weeks. There were 5 domains that could be described within SNOT-22, including nasal, ear, sleep, general and practical, and emotional; each domain was scored on a 5-category scale which ranged from 0: no problem to 5: problem as bad as it can be. The total score was the sum of response to each of the 22 questions and ranged from 0 (no disease) to 110 (worst disease), higher scores indicated worse HRQoL. Baseline was defined as the last available value before randomization.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
score on a scale | -11.58 (3.14) | -21.10 (3.14)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0104, ANCOVA; Least square mean difference = -9.52, 95% CI 2-sided [-16.81 to -2.24] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Received Systemic Corticosteroid (SCS) or Underwent Nasal Polyposis (NP) Surgery During the Study Treatment
Description: SCS for rescue treatment of nasal polyps or for another reason were prescribed to the participant by the site. For participants who had a surgery or had a scheduled date for surgery for NP, the reason (worsening signs and/or symptoms during the study), the expected or actual surgery date, the type and outcome of surgery was recorded in a specific e-case report form page. Percentage of participants who received SCS or underwent NP surgery during the study treatment are presented.
Time Frame: From randomization (Day 1) up to last dose of study treatment + 14 days, a maximum of 168 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
percentage of participants | 9.4 | 0

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment-Emergent Adverse Events Leading to Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment + 98 days, a maximum of 252 days
Population: The safety population included all participants randomly assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 32 | 31
Participants
  TEAEs | 20 | 23
  TESAEs | 0 | 4
  TEAEs leading to treatment discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs, SAEs and all-cause mortality (deaths) were collected from first dose of study treatment (Day 1) up to last dose of study treatment + 98 days, a maximum of 252 days
Description: Analysis was performed on the safety population.
Arm/Group | Placebo | Dupilumab 300 mg q2w
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 4/31
Other Adverse Events (participants affected / at risk) | 11/32 | 15/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Dupilumab 300 mg q2w (N=31)
Helicobacter Gastritis (Infections and infestations) | 0 (0) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Dupilumab 300 mg q2w (N=31)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (7) | 4 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Influenza Like Illness (General disorders) | 1 (1) | 2 (3)
Injection Site Reaction (General disorders) | 0 (0) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT05878093/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05878093/SAP_001.pdf